CLINICAL TRIAL: NCT03978104
Title: Impact of Okara and Bio-okara Food Product on Gut and Glycaemic Health in Middle-aged and Older Adults in Singapore
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: S4
Record Dates: First submitted 2019-05-24; First posted 2019-06-06 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Microbiota; Gastrointestinal Microbiome; Blood Glucose; Aging
Keywords: Okara; Soybean pulp; Soybean; Fibre; Gut microbiome; Microbiota; Gastrointestinal microbiome; Glycemic; Glycaemic; Middle-aged and older adults; Singapore

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Primary investigator of the study will be blinded in this intervention trial through blinding of the intervention allocation to subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Okara biscuits (Experimental): Subjects will consume their habitual diet with daily okara biscuit consumption accounting to 20 grams/ day of dry okara powder for 21 days.
  Interventions: Dietary Supplement: Okara biscuits
- Bio-okara biscuits (Experimental): Subjects will consume their habitual diet with daily bio-okara biscuit consumption accounting to 20 grams/ day of dry bio-okara powder for 21 days.
  Interventions: Dietary Supplement: Bio-okara biscuits
- Control biscuits (Experimental): Subjects will consume their habitual diet with daily control biscuit consumption for 21 days.
  Interventions: Dietary Supplement: Control biscuits

INTERVENTIONS:
Dietary Supplement: Okara biscuits — Consumption of okara-enriched biscuits together with habitual diet.
  Arms: Okara biscuits
Dietary Supplement: Bio-okara biscuits — Consumption of bio-okara-enriched biscuits together with habitual diet. Bio-okara is a form of fermented okara.
  Other Names: Fermented okara biscuits
  Arms: Bio-okara biscuits
Dietary Supplement: Control biscuits — Consumption of control biscuits together with habitual diet.
  Arms: Control biscuits

SUMMARY:
This research project aims to provide the scientific findings about the beneficial effects of okara (soybean pulp) consumption on gut and glycaemic health in middle-aged and older individuals in Singapore. In addition, it aims to examine the health promoting impact of bio-transformed okara in this population. We hypothesise that consuming a habitual diet with an okara (untreated or bio-transformed) incorporated food product will improve the gut microbiome composition and will increase the production of short chain fatty acids when compared to a same diet with no okara. Okara-based food product can also improve the glycaemic response in individuals compared to a product without okara in meal tolerance test (acute).

DETAILED DESCRIPTION:
For this double-blind, randomized, crossover experiment, the participants will complete a 16-week study period. Following a 1-wk pre-intervention baseline period, each participant will be randomly assigned to consume their habitual diet that either contains or do not contain okara food product (untreated and bio-transformed okara) for 3 weeks. The food product will be equivalent to a consumption of 20 g of okara (dried) per day. Following a 3-week dietary 'washout' period, the participants will be assigned to consume the other diets for another 3 weeks. This process will be repeated until each participant have completed all three interventions. Fecal and fasting-state blood samples will be obtained at study weeks 1, 4, 7, 10, 13, and 16, which correspond to before and end of the three 3-week intervention periods.

Additionally, during Weeks 1, 7 and 13, fasted participants will also be required to undergo a meal tolerance test. A cannula will first be inserted into the participant's forearm for blood sampling by a trained phlebotomist. One of three meals prepared by designated study personnel will then be randomly assigned during each visit, namely, control biscuit, untreated okara biscuit and bio-transformed okara biscuit. During each test, the participants will eat the prepared meal within 10 minutes and have blood samples drawn by intravenous cannulation at time = 0, 15, 30, 45, 60, 90, 120, 180 and 240 min, with time 0 being the time the participants first start eating the biscuits. The blood samples will analyzed for the postprandial blood glucose, insulin responses and lipid levels.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give an informed consent
2. Age 50 to 75 years
3. Willing to follow the study procedures

Exclusion Criteria:

All subjects meeting any of the exclusion criteria at baseline will be excluded from participation

1. Significant change in weight (≥ 3 kg body weight) during the past 3 months
2. Allergy to soy-based products
3. Acute illness at the study baseline
4. Exercising vigorously over the past 3 months
5. Following any restricted diet (e.g. vegetarian)
6. Smoking
7. Have a daily intake of more than 2 alcoholic drinks per day
8. Prescribed and taking antihypertensive/cholesterol-lowering/ type-2 diabetic medication which started less than 5 years prior to the intervention participation
9. Taking dietary supplements which may impact the outcome of interests (e.g. vitamin supplements, probiotic supplement etc.)
10. Pregnant, lactating, or planning pregnancy in the next 6 months
11. Insufficient venous access to allow the blood collection
12. Very high intake of fibre/ vegetables on a daily basis

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiome composition before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Gut microbiome composition will be determined via fecal samples of subjects at baseline and after each intervention period.
Change in fecal short chain fatty acids (SCFA) before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  SCFA will be determined via fecal samples of subjects at baseline and after each intervention period.
Change in serum short chain fatty acids (SCFA) before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  SCFA will be determined via serum samples of subjects at baseline and after each intervention period.
Change in fecal bile acids before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Bile acids will be determined via serum samples of subjects at baseline and after each intervention period.
Change in serum zonulin before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Serum zonulin will be determined via serum samples of subjects at baseline and after each intervention period.
Change in blood glucose levels before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Glucose levels will be determined via fasted blood samples of subjects at baseline and after each intervention period.
Change in blood insulin levels before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Insulin levels will be determined via fasted blood samples of subjects at baseline and after each intervention period.
Change in blood triglyceride levels before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Total triglyceride levels will be determined via fasted blood samples of subjects at baseline and after each intervention period.
Change in blood cholesterol levels before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Total cholesterol levels will be determined via fasted blood samples of subjects at baseline and after each intervention period.
Change in blood low-density lipoprotein-cholesterol levels before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  Low-density lipoprotein-cholesterol levels will be determined via fasted blood samples of subjects at baseline and after each intervention period.
Change in blood high-density lipoprotein-cholesterol levels before and after a 3 week intervention. | Baseline and post-intervention (at 3 weeks)
  High-density lipoprotein-cholesterol levels will be determined via fasted blood samples of subjects at baseline and after each intervention period.
Change in blood glucose levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Glucose levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood insulin levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Insulin levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood short-chain fatty acids levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Short-chain fatty acids levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood amino acid levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Amino acid levels will be determined via fasted blood samples of subjects and after consumption of intervention

SECONDARY OUTCOMES:
Change in blood pressure | Baseline and post-intervention (at 3 weeks)
  Blood pressure
Change in anthropometric measurements | Baseline and post-intervention (at 3 weeks)
  Waist circumference
Change in anthropometric measurements | Baseline and post-intervention (at 3 weeks)
  Weight
Change in anthropometric measurements | Baseline
  Height
Dietary assessment | Baseline and post-intervention (at 3 weeks)
  Dietary questionnaires (3-day food record)
Stool assessment | Baseline and post-intervention (at 3 weeks)
  Stool sampling questionnaire will be completed by subjects, which notes down food or alcohol consumed over the past 24 hours prior to collection, any discomfort, pain or bloating, flatulence, noticable changes in stool frequency or consistency, any blood in stool and any type of medication consumed over the past 3 months.
Stool assessment | Baseline and post-intervention (at 3 weeks)
  Bristol stool chart (Ranging from Type 1 to Type 7, with Type 3 or 4 being ideal.
Sleep quality assessment | Baseline and post-intervention (at 3 weeks)
  Pittsburgh sleep quality index questionnaire, with 7 different components assessing sleep and each component making up a minimum or 0 and maximum of 3 points. The full scale ranges from 0 to 21, with a lower score indicative of a better quality of sleep.
Sleep quality assessment | Baseline and post-intervention (at 3 weeks)
  Sleep evaluation questionnaire (survey) to assess eligibility for studies with sleep involved
Cognitive assessment | Baseline and post-intervention (at 3 weeks)
  Montreal cognitive assessment
Appetite assessment | Baseline and post-intervention (at 3 weeks)
  Visual analogue scale, with unit of measure being units on a scale
Change in blood amino acids levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Amino acid levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood triglyceride levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Total triglyceride levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood cholesterol levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Total cholesterol levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood low-density lipoprotein-cholesterol levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  Low-density lipoprotein-cholesterol levels will be determined via fasted blood samples of subjects and after consumption of intervention
Change in blood high-density lipoprotein-cholesterol levels over acute trial period | Time 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes held on pre- intervention arm visit (Every 6 weeks, up to 12 weeks).
  High-density lipoprotein-cholesterol levels will be determined via fasted blood samples of subjects and after consumption of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Principal Investigator — National University of Singapore
Locations (1):
- Department of Food Science and Technology; National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic data with any identifiable participant information will be de-identified prior to statistical analysis.

REFERENCES:
- [Background] Vong, W.C., X.Y. Hua, and S.-Q. Liu, Solid-state fermentation with Rhizopus oligosporus and Yarrowia lipolytica improved nutritional and flavour properties of okara. Lwt, 2018. 90: p. 316-322.
- [Background] Yogo, T., et al., Influence of Dried Okara-Tempeh on the Composition and Metabolites of Fecal Microbiota in Dogs. International Journal of Applied Research in Veterinary Medicine, 2011. 9(2): p. 176-183.
- [Background] Jimenez-Escrig A, Tenorio MD, Espinosa-Martos I, Ruperez P. Health-promoting effects of a dietary fiber concentrate from the soybean byproduct okara in rats. J Agric Food Chem. 2008 Aug 27;56(16):7495-501. doi: 10.1021/jf800792y. Epub 2008 Jul 18. PMID 18636739
- [Background] Lu, F., Y. Liu, and B. Li, Okara dietary fiber and hypoglycemic effect of okara foods. Bioactive Carbohydrates and Dietary Fibre, 2013. 2(2): p. 126-132.
- [Derived] Lee DPS, Gan AX, Sutanto CN, Toh KQX, Khoo CM, Kim JE. Postprandial glycemic and circulating SCFA concentrations following okara- and biovalorized okara-containing biscuit consumption in middle-aged and older adults: a crossover randomized controlled trial. Food Funct. 2022 Sep 22;13(18):9687-9699. doi: 10.1039/d2fo00526c. PMID 36040444